CLINICAL TRIAL: NCT05125991
Title: Evaluation of the Effectiveness of the Prepectoral Breast Reconstruction With Braxon Dermal Matrix: a Randomized Controlled Study
Brief Title: Evaluation of the Effectiveness of Prepectoral Breast Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IEO 1002/
Record Dates: First submitted 2021-10-25; First posted 2021-11-18 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prepectoral reconstruction (Experimental): Prepectoral breast reconstruction with Braxon dermal matrix
  Interventions: Procedure: Prepectoral reconstruction
- Submuscular reconstruction (Active Comparator): Submuscolar breast reconstruction
  Interventions: Procedure: Submuscolar reconstruction

INTERVENTIONS:
Procedure: Prepectoral reconstruction — Prepectoral breast reconstruction
  Arms: Prepectoral reconstruction
Procedure: Submuscolar reconstruction — Submuscolar breast reconstruction
  Arms: Submuscular reconstruction

SUMMARY:
The study plans to compare conventional submuscular reconstruction with definitive implant and muscle sparing reconstruction with definitive implant in selected patients. The two techniques are compared in terms of patient quality of life and satisfaction; patient related outcomes, reconstruction morbidity, early and late complications are also investigated.

DETAILED DESCRIPTION:
The study plans to compare conventional submuscular reconstruction with definitive implant and muscle sparing reconstruction with definitive implant in selected patients. The two techniques are compared in terms of patient quality of life and satisfaction; patient related outcomes, reconstruction morbidity, early and late complications are also investigated.

The study plans to collect robust data to support the prepectoral implant placement and complete coverage of implant with acellular dermal matrix in the clinical practice.

Consequently, the project plans to move toward evidence-based medicine in breast reconstruction, avoiding marketing influences and surgeon experience as the sole source of evidence.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent
2. Not smokers
3. No vascular comorbidities (diabetic, vasculitis, coagulation disorders)
4. BMI<30
5. CUP B-C (or mastectomy estimated weight less than 550gm)
6. Good subcutaneous layer (>1cm on pinch test measured in upper/medial quadrant)
7. No previous breast surgery
8. No previous breast irradiation
9. Breast Ptosis 1-2 according to Renault's classification
10. DCIS tumors
11. T1 T2 pN0 breast tumor with known favourable biologic features

Exclusion Criteria:

1. Impossibility of immediate reconstruction with definitive implants due to inadequacy of mastectomy flaps (inadequate in quantity and/or quality)
2. Positive sentinel node biopsy requiring complete axillary dissection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2019-09-03 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Satisfaction assessed by the BREAST-Q | 1 year
  The BREAST-Q survey is used to detect differences in patient satisfaction among the groups

SECONDARY OUTCOMES:
Immediate complications rate | 1 month
  Compare post operative complications
Short term complications rate | 6 months
  Compare short term post operative complications
Long term complications rate | 24 months
  Compare long term post operative complications
Percentage of capsular contracture | 1 year
  Compare overall aesthetic outcomes (percentage of capsular contracture) using standardized photographs assessed by independent blinded observers

CONTACTS AND LOCATIONS:
Overall Officials: Francesca De Lorenzi, PhD, MD, Principal Investigator — European Institute of Oncology; Paolo Veronesi, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy

IPD SHARING:
Plan to Share IPD: No